CLINICAL TRIAL: NCT05902637
Title: The Efficacy of Mapping for Cognitive Prostate Biopsy: a Prospective, Randomized Study
Brief Title: The Efficacy of Mapping for Cognitive Prostate Biopsy
Acronym: MAPROSTATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tarik Emre Sener, Associating Professor, MD, Marmara University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MAR.UAD.006
Record Dates: First submitted 2023-03-17; First posted 2023-06-15 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostatic Neoplasms; Prostate Disease; Prostate Cancer Stage
Keywords: Prostate; Cancer; Mapping; Genitourinary Radiology; Transrectal; Biopsy; Rectal examination; Method; Efficacy; Prostate mapping; Cognitive; prospective; Randomized
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases; Neoplasms | interventions — Microtubule-Associated Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prostate Mapping Used (Active Comparator): Those patients' Multiparametric Prostate Magnetic Resonance (MPMR) imaging's have been assessed by a genitourinary radiologist to guide the surgeon who performs cognitive prostate biopsy
  Interventions: Procedure: Performing cognitive prostate biopsy with a radiologist's guidance with map
- Prostate Mapping not Used (Sham Comparator): Those patients' Multiparametric Prostate Magnetic Resonance (MPMR) imaging's have not been assessed by a genitourinary radiologist to guide the surgeon who performs cognitive prostate biopsy. Surgeon assesses the Multiparametric Prostate Magnetic Resonance (MPMR) imaging's by him/herself
  Interventions: Procedure: Performing cognitive prostate biopsy without a radiologist's guidance with map

INTERVENTIONS:
Procedure: Performing cognitive prostate biopsy with a radiologist's guidance with map — All patients will undergo prostate biopsy under local or general anesthesia with transrectal ultrasonography by a single surgeon after mapping extracted by a single genitourinary radiologist in the Department of Radiology of our hospital.
  Arms: Prostate Mapping Used
Procedure: Performing cognitive prostate biopsy without a radiologist's guidance with map — All patients will undergo cognitive prostate biopsy under local or general anesthesia with transrectal ultrasonography by a single surgeon after reported by a single genitourinary radiologist in the Department of Radiology of our hospital.
  Arms: Prostate Mapping not Used

SUMMARY:
Today, many centers still perform Magnetic Resonance Imaging (MRI) cognitive prostate biopsy. The efficacy of detecting clinically significant prostate cancer, which is thought to be due to the experience of the urologist who performed the sampling and the difference in experience of the radiologists who performed the Multiparametric Prostate Magnetic Resonance (MPMR) evaluation, has been reported between 25% and 34% in the literature.

In order to eliminate this reporting and sampling difference, The goal of this interventional study is to compare the effectiveness of Multiparametric Prostate Magnetic Resonance (MPMR) Imaging routinely taken before biopsy with a single-center randomized and prospective study and prostate biopsies to be performed by the same urologist with the mapping technique created by a single genitourinary radiologist working in our center with standard cognitive prostate biopsy and to contribute to the literature Type of study: Clinical trial participant population: Male patients with elevated serum Prostate Specific Antigen (PSA) or indicated prostate biopsy by Magnetic Resonance Imaging (MRI) imaging and underwent Multiparametric Prostate Magnetic Resonance (MPMR) before the procedure Participants will undergo transrectal prostate biopsy with or without mapping, Researches will compare to see if the cancer detection rates differ

DETAILED DESCRIPTION:
In this preliminary clinical study, 200 patients who underwent cognitive prostate biopsy under the guidance of transrectal ultrasonography between 01.03.2023 and 01.09.2023 by Marmara University Department of Urology, Department of Urooncology due to serum Prostate Specific Antigen (PSA) elevation and/or abnormal rectal examination findings will be included in the study. All patients will undergo prostate biopsy under local or general anesthesia with transrectal ultrasonography by a single surgeon after mapping or report is extracted by a single genitourinary radiologist in the Department of Radiology of our hospital.

In the power analysis, 200 patients were included in the study with the prediction that the efficacy difference would be calculated as 5%. All patients will be randomized to two equal groups by the flip-flip method.

1. Multiparametric Prostate Magnetic Resonance Imaging and reports of the mapped patients will be examined and cognitive prostate biopsy will be performed by looking at the map (Sample Figure 1,2) created by the same urologist and the same radiologist (Sample Figure 1,2). Standard 12 core (6 peripheral zones from both lobes) will be sampled and 4 extra biopsies will be taken from Prostate Imaging-Reporting and Data System (PI-RADS) Category 3-4-5 areas in the mapping.
2. Based on the Multiparametric Prostate Magnetic Resonance Imaging reports and images, without mapping by the radiologist, only the standard 12 core (6 from each peripheral zone from both lobes) determined cognitively by the urologist and 4 extra biopsies from the Prostate Imaging-Reporting and Data System (PI-RADS) Category 3-4-5 areas described in the report will be taken.

And then the biopsy results will be compared to see the efficacy of mapping

ELIGIBILITY:
Inclusion Criteria:

* Patients with elevated serum Prostate Specific Antigen (PSA)
* Indicated prostate biopsy by MR imaging and underwent Multiparametric Prostate Magnetic Resonance (MPMR) imaging before the procedure

Exclusion Criteria:

* Patients with suspicious Rectal Examination findings
* Patients who cannot enter Multiparametric Prostate Magnetic Resonance (MPMR) imaging for various reasons (such as Multiparametric Prostate Magnetic Resonance (MPMR) imaging incompatible pacemaker, Chronic Kidney Disease)
* Patients with diagnosed prostate cancer and active surveillance
* Patients without indication for prostate biopsy
* Patients with very high serum Prostate Specific Antigen (PSA) levels (>15)
* Patients who are planned to start treatment by diagnosing with standard 12 core biopsy without losing time with imaging method
* Patients who do not want to participate in the study.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 175 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Detecting prostate cancer | 6 months
  Detection of any kind or any grade of prostate cancer on the pathological specimen of Transrectal Ultrasound Guided Prostate Biopsy:
  * Detection of prostate adenocarcinoma of any ISUP (grade 1, grade 2, grade 3, grade 4 or grade 5) / Gleason score (Gleason score 6-10)
  * Detection of non-adenocarcinoma cancers of prostate (small cell carcinoma, neuroendocrine tumor, sarcomatous carcinoma, signet ring cell, basaloid carcinoma, pseudohyperplastic carcinoma, lymphoepithelioma-like carcinoma, adenosquamous cell carcinoma)

CONTACTS AND LOCATIONS:
Overall Officials: Haydar Kamil Cam, Prof., Study Chair — Marmara University, School of Medicine, Department of Urology
Locations (1):
- Marmara University, School of Medicine, Department of Urology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Culp MB, Soerjomataram I, Efstathiou JA, Bray F, Jemal A. Recent Global Patterns in Prostate Cancer Incidence and Mortality Rates. Eur Urol. 2020 Jan;77(1):38-52. doi: 10.1016/j.eururo.2019.08.005. Epub 2019 Sep 5. PMID 31493960
- [Background] Bell KJ, Del Mar C, Wright G, Dickinson J, Glasziou P. Prevalence of incidental prostate cancer: A systematic review of autopsy studies. Int J Cancer. 2015 Oct 1;137(7):1749-57. doi: 10.1002/ijc.29538. Epub 2015 Apr 21. PMID 25821151
- [Background] Jansson KF, Akre O, Garmo H, Bill-Axelson A, Adolfsson J, Stattin P, Bratt O. Concordance of tumor differentiation among brothers with prostate cancer. Eur Urol. 2012 Oct;62(4):656-61. doi: 10.1016/j.eururo.2012.02.032. Epub 2012 Feb 24. PMID 22386193
- [Background] Lendinez-Cano G, Ojeda-Claro AV, Gomez-Gomez E, Morales Jimenez P, Flores Martin J, Dominguez JF, Amores J, Cozar JM, Bachiller J, Juarez A, Linares R, Garcia Galisteo E, Alvarez Ossorio JL, Requena Tapia MJ, Moreno Jimenez J, Medina Lopez RA; AEU-PIEM/2018/000 Investigators. Prospective study of diagnostic accuracy in the detection of high-grade prostate cancer in biopsy-naive patients with clinical suspicion of prostate cancer who underwent the Select MDx test. Prostate. 2021 Sep;81(12):857-865. doi: 10.1002/pros.24182. Epub 2021 Jun 29. PMID 34184761
- [Background] Oerther B, Engel H, Bamberg F, Sigle A, Gratzke C, Benndorf M. Cancer detection rates of the PI-RADSv2.1 assessment categories: systematic review and meta-analysis on lesion level and patient level. Prostate Cancer Prostatic Dis. 2022 Feb;25(2):256-263. doi: 10.1038/s41391-021-00417-1. Epub 2021 Jul 6. PMID 34230616
- [Background] Barkovich EJ, Shankar PR, Westphalen AC. A Systematic Review of the Existing Prostate Imaging Reporting and Data System Version 2 (PI-RADSv2) Literature and Subset Meta-Analysis of PI-RADSv2 Categories Stratified by Gleason Scores. AJR Am J Roentgenol. 2019 Apr;212(4):847-854. doi: 10.2214/AJR.18.20571. Epub 2019 Feb 26. PMID 30807218
- [Background] Presti JC Jr. Prostate biopsy: how many cores are enough? Urol Oncol. 2003 Mar-Apr;21(2):135-40. doi: 10.1016/s1078-1439(03)00006-1. PMID 12856642
- [Background] Wegelin O, Exterkate L, van der Leest M, Kummer JA, Vreuls W, de Bruin PC, Bosch JLHR, Barentsz JO, Somford DM, van Melick HHE. The FUTURE Trial: A Multicenter Randomised Controlled Trial on Target Biopsy Techniques Based on Magnetic Resonance Imaging in the Diagnosis of Prostate Cancer in Patients with Prior Negative Biopsies. Eur Urol. 2019 Apr;75(4):582-590. doi: 10.1016/j.eururo.2018.11.040. Epub 2018 Dec 3. PMID 30522912